CLINICAL TRIAL: NCT02192814
Title: A Multicenter, Open-label Study to Evaluate the Safety and Tolerability of Intravenous Lacosamide as Replacement for Oral Lacosamide in Japanese Adults With Partial-onset Seizures With or Without Secondary Generalization
Brief Title: Open-label Study to Evaluate the Safety and Tolerability of iv Lacosamide in Japanese Adults With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0024; EP0024 (Other: JAPIC)
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Results first posted 2015-12-04 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy; Partial-onset Seizures
Keywords: Lacosamide; LCM; Epilepsy; Partial-onset seizures; iv
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (LCM) (Experimental): On Day - 1, LCM oral tablets were administered in accordance with each subject's LCM dosage regimen in EP0009 (NCT01832038). The oral tablets were taken from EP0009 supply.
  During the Treatment Period, subjects received a 30-minute infusion of intravenous (iv) LCM twice daily, once in the morning and once in the evening, for 5 days.
  The daily dose of iv LCM was the same as the subject's daily dose of oral LCM in EP0009 (200 - 400 mg/day).
  Interventions: Drug: Lacosamide (200 mg/20 mL)

INTERVENTIONS:
Drug: Lacosamide (200 mg/20 mL) — Active Substance: Lacosamide
  Pharmaceutical form: Solution for intravenous (iv) infusion
  Concentration: adapted on concentration of oral dose in EP0009
  Route of Administration: Drip infusion
  Other Names: Vimpat

SUMMARY:
EP0024 is a Phase 3, multicenter, open-label study to evaluate the safety and tolerability of intravenous (iv) lacosamide (LCM). Adjunctive iv LCM therapy (200 mg/day to 400 mg/day) will be administered for 5 days as replacement for oral LCM tablets in Japanese adults with partial-onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese and enrolled in EP0009 (NCT01832038) receiving oral Lacosamide (LCM) for the treatment of partial-onset seizures and has been enrolled for at least 8 weeks
* Subject has been on a stable twice daily (bid) dosage regimen of LCM 200 mg/ day to 400 mg/ day, for the 2 weeks prior to entry into EP0024
* Subject has been receiving no more than 3 concomitant Antiepileptic Drugs (AEDs) at doses that have remained stable for the 2 weeks prior to entry into EP0024

Exclusion Criteria:

* Subject has a history of any kind of status epilepticus within 12-month period prior to study entry
* Subject has actual suicidal ideation as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Since Last Visit" version of the Columbia-Suicide Severity Rating Scale (C-SSRS)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1-877-822-9493
Locations (5):
- Japan (5):
  - 81027, Hamamatsu
  - 81024, Kodaira
  - 81025, Sapporo
  - 81003, Shizuoka
  - 81023, Suita

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, open-label study started recruiting in June 2014.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS), consisting of all enrolled subjects who received at least 1 infusion of iv LCM.
Groups:
- Lacosamide (LCM): On Day - 1, Lacosamide (LCM) oral tablets were administered in accordance with each subject's LCM dosage regimen in EP0009 (NCT01832038). The oral tablets were taken from EP0009 supply.
  During the Treatment Period, subjects received a 30-minute infusion of intravenous (iv) LCM twice daily, once in the morning and once in the evening, for 5 days.
  The daily dose of iv LCM was the same as the subject's daily dose of oral LCM in EP0009 (200 - 400 mg/day).
Period: Overall Study
Arm/Group | Lacosamide (LCM)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participant Flow refers to the Safety Set (SS), consisting of all enrolled subjects who received at least 1 infusion of iv LCM.
  Subjects participating in EP0009 (NCT01832038) have been enrolled to EP0024.
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 55.99 (13.13)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.07 (8.63)

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of Subjects Experiencing at Least One Adverse Event During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: During the study (Screening through End of Study (Day -1 through Day 6))
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Number; unit: participants
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
participants | 4

2. Primary Outcome: The Total Number of Subject Withdrawal Due to Adverse Events During the Study
Description: as for outcome 1
Time Frame: During the study (Screening through End of Study (Day -1 through Day 6))
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Number; unit: participants
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
participants | 0

3. Secondary Outcome: Plasma Trough Concentration (Ctrough) for Lacosamide (LCM) on Day 1
Time Frame: 20 minutes prior infusion at Day 1
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 4.738 (50.5)

4. Secondary Outcome: Plasma Trough Concentration (Ctrough) for Lacosamide (LCM) on Day 2
Time Frame: 20 minutes prior infusion at Day 2
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 4.004 (55.4)

5. Secondary Outcome: Plasma Trough Concentration (Ctrough) for Lacosamide (LCM) on Day 5
Time Frame: 20 minutes prior infusion at Day 5
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 3.615 (60.0)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Lacosamide (LCM) (End of Infusion) on Day 1
Time Frame: 20 minutes prior infusion at Day 1
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 10.838 (46.6)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Lacosamide (LCM) (End of Infusion) on Day 2
Time Frame: 20 minutes prior infusion at Day 2
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 10.330 (50.0)

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Lacosamide (LCM) (End of Infusion) on Day 5
Time Frame: 20 minutes prior infusion at Day 5
Population: The Safety Set (SS) consisted of all enrolled subjects who received at least 1 infusion of iv LCM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lacosamide (LCM)
Number analyzed (Participants) | 9
µg/mL | 9.621 (38.8)

9. Other Pre Specified Outcome: The Cumulative Partial-onset Seizure Frequency From Day -1 to Day 5
Description: No descriptive statistics have been calculated for this exploratory Outcome Measure.
Time Frame: From Day -1 to Day 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Screening Period (Day -1) until End-of-Study Period (Day 6).
Description: Adverse Events refer to the Safety Set (SS) which constisted of all all enrolled subjects who received at least 1 infusion of iv LCM.
Groups:
- Lacosamide (LCM): On Day - 1, Lacosamide (LCM) oral tablets were administered in accordance with each subject's LCM dosage regimen in EP0009 (NCT01832038). The oral tablets were taken from EP0009 supply.
  During the Treatment Period, subjects received a 30-minute infusion of intravenous (iv) LCM twice daily, once in the morning and once in the evening, for 5 days.
  The daily dose of iv LCM was be the same as the subject's current daily dose of oral LCM in EP0009 (200 - 400 mg/day).
Arm/Group | Lacosamide (LCM)
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (LCM) (N=9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days